CLINICAL TRIAL: NCT03140176
Title: REAL-WORLD CLINICAL PATTERNS OF CARE AND OUTCOMES AMONG PATIENTS IN AFRICA MIDDLE EAST (AFME) WITH METASTATIC RENAL CELL CARCINOMA (MRCC) RECEIVING SUNITINIB AS FIRST LINE THERAPY (OPTIMISE).
Brief Title: Real-world Clinical Patterns Of Care And Outcomes Among AfME mRCC Patients Receiving Sunitinib as First Line Therapy.
Acronym: OPTIMISE
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early due to the inability to recruit the planned number of patients
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181223
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Sunitinib; Metastatic Renal Cell Carcinoma; Africa Middle East
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sunitinib — Sunitinib is an FDA approved targeted therapy for use as first line therapy for patients with metastatic renal cell carcinoma.
  Other Names: Sutent

SUMMARY:
OPTIMISE is designed to provide knowledge regarding the use of Sunitinib as 1st line treatment and 2nd line treatment selected (Sunitinib-different sequence) with respect to efficacy outcomes, adverse events, and health related QoL in the real life setting.

DETAILED DESCRIPTION:
OPTIMISE study objectives are dual and aim primarily to increase the knowledge regarding the outcomes from Sunitinib use on one hand; and outcomes from the combined Sunitinib-2nd line sequence on the other hand in real life clinical practice.

This will be addressed in many countries across AfME and in individual country cohorts to understand specificities and differences in use and outcomes

ELIGIBILITY:
* Inclusion Criteria:

  1. Patients being treated with SU as 1st line treatment according to the approved therapeutic indication.
  2. Histologically confirmed diagnosis of mRCC (clear cell RCC as well as nonclear cell RCC) with measurable disease according to RECIST 1.1
  3. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

     Exclusion Criteria:

  <!-- -->

  1. Patients being treated with cytokines or any other treatment other than SU in 1st line setting
  2. Patients presenting with a known hypersensitivity to SU or its metabolites will not be included in the study per the label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic renal cell carcinoma being treated with Sunitinib as the first line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Algeria (3):
  - Pierre Et Marie Curie Center, Algers
  - CAC Annaba, Annaba
  - Hanene Djedi, Annaba
- Egypt (3):
  - Kasr Al Aini, Cairo
  - National Cancer Institute, Cairo
  - Demerdash Hospital, Cairo
- Kuwait Cancer Control Center, Kuwait City, Kuwait
- Institut National D'Oncologie, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged 18 years and above diagnosed with advanced metastatic renal cell cancer (mRCC) and treated with sunitinib as first line treatment according to the approved therapeutic indication in real world practice were enrolled in this observational study. Participants were enrolled across Africa and Middle East (AfME) countries.
Pre-assignment Details: A total of 77 participants with advanced RCC were enrolled in the study, of which 3 participants were excluded from analysis as they were not eligible. Only 74 enrolled participants were eligible to be included in the analysis of the study. Data was collected in routine clinical practice and from medical records.
Groups:
- Sunitinib: Eligible participants diagnosed with mRCC, who on enrollment into the study, initiated treatment with sunitinib as first line treatment in real world clinical routine practice, were included. Data was collected in routine clinical practice and studied from medical records.
Period: Overall Study
Arm/Group | Sunitinib
Started | 74
Completed | 0
Not Completed | 74
Not completed — Reason missing | 23
Not completed — Death | 33
Not completed — Disease progression | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Population: Full analysis set included all eligible participants enrolled in the study, whatever the therapeutic strategy used during the observation period.
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black/ African Descent | 2
  Caucasian | 18
  Middle Eastern | 45
  Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from when the participant received the first dose of sunitinib to the time of progression or death due to any cause, which occurred first. The time of progression was the date of the first tumor assessment where the progression was notified as response to therapy, over the sunitinib treatment. Participants who discontinued the study for any reason, including unacceptable toxicity during the treatment period, who remained alive and without disease progression, were censored at the last disease assessment that verified lack of disease progression. As per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, disease progression was defined as at least a 20% increase (including an absolute increase of at least 5 millimeters [mm]) in the sum of the longest dimensions of the target lesions taking as a reference smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From date of first dose of sunitinib to date of progression or death or censored date, whichever occurred first (up to maximum of 36 months)
Population: Full analysis set included all eligible participants enrolled in the study, whatever the therapeutic strategy used during the observation period. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 70
Days | 321.0 [115.0 to 546.0]

2. Primary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from when the participant received the first dose of sunitinib to the time of sunitinib discontinuation (date completed by the physician). In case of death when the participant was still treated with sunitinib, date of death was considered as date of discontinuation. If no sunitinib discontinuation was reported during the follow-up visits, participants were censored to the last follow-up visit.
Time Frame: From date of first dose of sunitinib until the date of discontinuation or censored date (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Days | 348.0 [109.0 to 546.0]

3. Secondary Outcome: Objective Response Rate (ORR) at Months 3, 6, 9 and 12
Description: ORR was defined as the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.1. As per RECIST 1.1 criteria: CR = disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm. Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis); PR = at least 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters.
Time Frame: Months 3, 6, 9 and 12
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Percentage of participants
  Month 3 | 17.6
  Month 6 | 9.5
  Month 9 | 8.1
  Month 12 | 2.7

4. Secondary Outcome: Number of Participants With Recommended Starting Dose of Sunitinib
Description: The recommended starting dose of sunitinib was 50 milligrams (mg) per day, 4 weeks on treatment followed by 2 weeks off.
Time Frame: At initiation of sunitinib (Day 0)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants | 29

5. Secondary Outcome: Number of Participants With Other Starting Doses
Description: Number of participants with other starting doses of sunitinib (50 mg per day, 2 weeks on, 1 week off; 37.5 mg per day for 2 weeks on and 1 week off; 25 mg per day for 2 weeks on and 1 week off; 37.5 mg per day 4 weeks on and 2 weeks off) were reported in this outcome measure.
Time Frame: At initiation of sunitinib (Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 45
Participants
  50 mg per day, 2 weeks on, 1 week off | 41
  37.5 mg per day for 2 weeks on and 1 week off | 2
  25 mg per day for 2 weeks on and 1 week off | 1
  37.5 mg per day 4 weeks on and 2 weeks off | 1

6. Secondary Outcome: Number of Participants With Moderate Chronic Liver Failure, With 2 Milligrams (mg) Twice Daily (BID) as Starting Dose
Time Frame: At initiation of sunitinib (Day 0)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants | 0

7. Secondary Outcome: Average Dose Received Over the Sunitinib Treatment Period
Time Frame: During treatment period (up to 12 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Sunitinib
Number analyzed (Participants) | 67
Milligrams | 7917.1 (6834.5)

8. Secondary Outcome: Dose Intensity of Sunitinib
Description: Dose intensity was defined as defined as the sum of sunitinib daily doses divided by the duration of sunitinib treatment in days (delay between the first sunitinib dose and the last dose, including temporary interruption).
Time Frame: During treatment period (up to 12 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligrams per day
Arm/Group | Sunitinib
Number analyzed (Participants) | 67
Milligrams per day | 48.5 (5.1)

9. Secondary Outcome: Number of Participants With Change in Dose or Schedule of Sunitinib
Description: Number of participants with change in dose or schedule of sunitinib at the specified time points were reported in this outcome measure.
Time Frame: Month 3, 6, 9 and 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants
  Month 3 | 7
  Month 6 | 3
  Month 9 | 2
  Month 12 | 0

10. Secondary Outcome: Number of Participants With Dose Increase
Time Frame: During treatment period (up to 12 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants | 0

11. Secondary Outcome: Number of Participants With Temporary Interruption During the Sunitinib Treatment Period
Time Frame: During treatment period (up to 12 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants | 15

12. Secondary Outcome: Time to First Interruption
Time Frame: During treatment period (up to 12 months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 15
Days | 130.0 [49.0 to 252.0]

13. Secondary Outcome: Time to All Interruptions
Time Frame: During treatment period (up to 12 months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 15
Days | 109.0 [49.0 to 253.0]

14. Secondary Outcome: Number of Participants According to Reasons for Temporary Interruption
Description: Number of participants according to reasons for temporary interruption (adverse events, logistical, personal and intolerant to sunitinib) at specified time points is presented in this outcome measure.
Time Frame: Months 3, 6, 9 and 12
Population: Full analysis set included all eligible participants enrolled in the study, whatever the therapeutic strategy used during the observation period. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 15
Participants
  Month 3: number analyzed (Participants) | 8
  Month 3: Adverse events | 5
  Month 3: Logistical | 1
  Month 3: Personal | 1
  Month 3: Intolerant to Sunitinib | 1
  Month 6: number analyzed (Participants) | 3
  Month 6: Adverse events | 3
  Month 6: Logistical | 0
  Month 6: Personal | 0
  Month 6: Intolerant to Sunitinib | 0
  Month 9: number analyzed (Participants) | 1
  Month 9: Adverse events | 1
  Month 9: Logistical | 0
  Month 9: Personal | 0
  Month 9: Intolerant to Sunitinib | 0
  Month 12: number analyzed (Participants) | 3
  Month 12: Adverse events | 3
  Month 12: Logistical | 0
  Month 12: Personal | 0
  Month 12: Intolerant to Sunitinib | 0

15. Secondary Outcome: Number of Participants With Sunitinib Discontinuation
Description: Number of participants with sunitinib discontinuation at specified time points is presented in this outcome measure.
Time Frame: Months 3, 6, 9 and 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants
  Month 3 | 15
  Month 6 | 4
  Month 9 | 4
  Month 12 | 6

16. Secondary Outcome: Number of Participants According to Reasons for Sunitinib Discontinuation
Description: Number of participants according to reasons for sunitinib discontinuation (death, intolerability, progression) at specified time points is presented in this outcome measure.
Time Frame: Months 3, 6, 9 and 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 29
Participants
  Month 3: number analyzed (Participants) | 15
  Month 3: Death | 1
  Month 3: Intolerability | 4
  Month 3: Progression | 10
  Month 3: Unknown/Missing | 0
  Month 6: number analyzed (Participants) | 4
  Month 6: Death | 0
  Month 6: Intolerability | 1
  Month 6: Progression | 3
  Month 6: Unknown/Missing | 0
  Month 9: number analyzed (Participants) | 4
  Month 9: Death | 0
  Month 9: Intolerability | 1
  Month 9: Progression | 2
  Month 9: Unknown/Missing | 1
  Month 12: number analyzed (Participants) | 6
  Month 12: Death | 0
  Month 12: Intolerability | 1
  Month 12: Progression | 5
  Month 12: Unknown/Missing | 0

17. Secondary Outcome: Median Duration of Sunitinib Treatment
Description: Median duration of treatment was defined as the time between the sunitinib initiation and the sunitinib discontinuation date or the last follow-up date with sunitinib treatment.
Time Frame: From date of first dose of sunitinib until discontinuation or last follow-up date with sunitinib treatment (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Days | 169.5 [87.0 to 362.0]

18. Secondary Outcome: Combined Progression Free Survival
Description: Combined PFS was defined as the time from when the participants received the first dose of sunitinib as first line, until progression or death due to any cause while on the 2nd line treatment, whichever occurred first during the 2nd line sequence treatment. As per RECIST version 1.1, disease progression was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of the longest dimensions of the target lesions taking as a reference smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: From date of first dose of sunitinib until progression or death whichever occurred first during second line treatment (up to maximum of 36 months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 70
Days | 502.0 [215.0 to 660.0]

19. Secondary Outcome: Combined TTF for the Sunitinib-2nd Line Sequence
Description: Combined TTF was defined as the time from when the participant received the first dose with sunitinib as first line, to the time of 2nd line sequence discontinuation (date completed by the physician).
Time Frame: From date of first dose of sunitinib until discontinuation of second line treatment (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Days | 378.0 [146.0 to 793.0]

20. Secondary Outcome: Combined PFS According to Type of Second Line Treatment
Description: Combined PFS was defined as the time from when the participants received the first dose of sunitinib as first line, until progression or death due to any cause while on the 2nd line treatment, whichever occurred first during the 2nd line sequence treatment. As per RECIST version 1.1, disease progression was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of the longest dimensions of the target lesions taking as a reference smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions. Combined PFS according to the type of second line treatment (best supportive care [BSC], tyrosine kinase inhibitors [TKI] including pazopanib and mammalian target of rapamycin [mTOR] inhibitors including everolimus) were reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
Days
  BSC: number analyzed (Participants) | 13
  BSC | 169.0 [144.0 to 539.0]
  TKI: number analyzed (Participants) | 12
  TKI | 948.0 [435.0 to 1095.0]
  mTOR: number analyzed (Participants) | 3
  mTOR | 399.0 [215.0 to 399.0]

21. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of first sunitinib dose to the date of death of any cause.
Time Frame: From date of first dose of sunitinib to the date of death of any cause (up to maximum of 36 months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 70
Days | 544.0 [146.0 to 794.0]

22. Secondary Outcome: Number of Participants Experiencing At Least One Adverse Event (AE) of Any Grade
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. AEs were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) as follows: Grade 1: mild AE, Grade 2: moderate AE, Grade 3: severe AE, Grade 4: life-threatening consequences and urgent intervention indicated, Grade 5: death related to AE. In this outcome measure, number of participants with at least one AE of any grade is reported.
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants | 51

23. Secondary Outcome: Number of Most Common AEs of Any Grade by Preferred Term
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. AEs were graded according to NCI-CTCAE as follows: Grade 1: mild AE, Grade 2: moderate AE, Grade 3: severe AE, Grade 4: life-threatening consequences and urgent intervention indicated, Grade 5: death related to AE. In this outcome measure, number of most common AEs of any grade is presented. Only events captured as deaths (preferred term) are reported as deaths in the data table.
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Number; unit: Events
Units Other Than Participants: Adverse events
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Number analyzed (Adverse events) | 150
Events
  Death | 19
  Anemia | 8
  Diarrhea | 8
  Mucosal inflammation | 8
  Vomiting | 8

24. Secondary Outcome: Number of Events of Diarrhea, Hypertension, Fatigue, Asthenia, Palmar-plantar Erythrodysesthesia Syndrome, Nausea, Stomatitis, Neutropenia, Lymphopenia and Elevated Lipase
Description: Number of events of diarrhea, hypertension, fatigue, asthenia, palmar-plantar erythrodysesthesia syndrome, nausea, stomatitis, neutropenia, lymphopenia and elevated lipase were reported in this outcome measure.
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Number; unit: Events
Units Other Than Participants: Adverse events
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Number analyzed (Adverse events) | 150
Events
  Diarrhea | 8
  Hypertension | 2
  Fatigue | 4
  Asthenia | 4
  Palmar-plantar erythrodysesthesia syndrome | 6
  Nausea | 2
  Stomatitis | 3
  Neutropenia | 1
  Lymphopenia | 0
  Elevated lipase | 0

25. Secondary Outcome: Number of Participants With Serious Adverse Events and Non-Serious AEs
Description: A serious adverse event was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. In this outcome measure, number of participants with serious adverse events and non-serious adverse events are reported.
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants
  Serious adverse events | 35
  Non-serious AEs | 35

26. Secondary Outcome: Number of Adverse Events According to Grade
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. AEs were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) as follows: Grade 1: mild AE, Grade 2: moderate AE, Grade 3: severe AE, Grade 4: life-threatening consequences and urgent intervention indicated, Grade 5: death related to AE.
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Number; unit: Events
Units Other Than Participants: Adverse events
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Number analyzed (Adverse events) | 150
Events
  Grade 1 | 35
  Grade 2 | 38
  Grade 3 | 32
  Grade 4 | 23
  Grade 5 | 22

27. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to AEs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage. In this outcome measure, number of participants who discontinued treatment due to AEs are reported.
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants | 20

28. Secondary Outcome: Duration of Treatment Until Discontinuation for AEs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product. The event need not necessarily have a causal relationship with the product treatment or usage.
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 20
Days | 572 [201 to 1079]

29. Secondary Outcome: Number of Participants Who Died Due to Any Cause
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 74
Participants | 33

30. Secondary Outcome: Number of Participants According to the Cause of Death
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 33
Participants
  Other cause | 11
  Tumor-related | 22

31. Secondary Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index-19 (FKSI-19) Total Scores
Description: The FKSI-19 is a disease-specific instrument that assessed symptoms of importance in renal cancer participants. It consisted of 4 subscales (FKSI-Disease Related Symptoms [DRS]-Physical [P]-12 items, FKSI-DRS-Emotional [E]-1 item, treatment side effects [TSE]-3 items, functional wellbeing [FWB]-3 items). Participants were required to respond to a total of 19 questions regarding symptoms, side effects and wellbeing on a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The total FKSI scores were calculated as the sum of the item responses divided by the number of items completed multiplied by the total number of items in the scale and ranged from 0 (severely symptomatic) to 76 (asymptomatic), where higher scores indicated better health.
Time Frame: Day 0, Month 3, 6, 9, 12, 18 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 68
Units on a scale
  Day 0 | 50.6 (12.4)
  Month 3: number analyzed (Participants) | 58
  Month 3 | 49.8 (13.9)
  Month 6: number analyzed (Participants) | 32
  Month 6 | 56.1 (11.0)
  Month 9: number analyzed (Participants) | 26
  Month 9 | 51.6 (14.5)
  Month 12: number analyzed (Participants) | 16
  Month 12 | 54.1 (15.4)
  Month 18: number analyzed (Participants) | 11
  Month 18 | 53.3 (9.4)
  Month 24: number analyzed (Participants) | 5
  Month 24 | 55.2 (9.6)

32. Secondary Outcome: Functional Assessment of Cancer Therapy Kidney Symptom Index-19 (FKSI-19) Sub-scale Scores
Description: The FKSI-19 is a disease-specific instrument that assessed symptoms of importance in renal cancer participants. It consisted of 4 subscales (FKSI-DRS-P: 12 items, FKSI-DRS-E: 1 item, TSE: 3 items, FWB: 3 items). Participants were required to respond to the items in each subscale on a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The FKSI subscale scores were calculated as the sum of item responses divided by the number of items completed multiplied by the total number of items in the subscale and ranged from 0 (severely symptomatic) to 48 (asymptomatic) for FKSI-DRS-P, 0 (severely symptomatic) to 4 (asymptomatic) for FKSI-DRS-E and 0 (severely symptomatic) to 12 (asymptomatic) for TSE and FWB; higher scores indicated better health.
Time Frame: Day 0, Month 3, 6, 9, 12, 18 and 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 68
Units on a scale
  FKSI-DRS-P; Day 0 | 31.9 (8.8)
  FKSI-DRS-P; Month 3: number analyzed (Participants) | 58
  FKSI-DRS-P; Month 3 | 33.2 (9.1)
  FKSI-DRS-P; Month 6: number analyzed (Participants) | 32
  FKSI-DRS-P; Month 6 | 37.6 (7.1)
  FKSI-DRS-P; Month 9: number analyzed (Participants) | 26
  FKSI-DRS-P; Month 9 | 34.7 (8.9)
  FKSI-DRS-P; Month 12: number analyzed (Participants) | 16
  FKSI-DRS-P; Month 12 | 35.6 (9.2)
  FKSI-DRS-P; Month 18: number analyzed (Participants) | 11
  FKSI-DRS-P; Month 18 | 34.6 (6.3)
  FKSI-DRS-P; Month 24: number analyzed (Participants) | 5
  FKSI-DRS-P; Month 24 | 37 (6.6)
  FKSI-TSE; Day 0 | 10.3 (1.6)
  FKSI-TSE; Month 3: number analyzed (Participants) | 58
  FKSI-TSE; Month 3 | 9.6 (2.1)
  FKSI-TSE; Month 6: number analyzed (Participants) | 32
  FKSI-TSE; Month 6 | 9.8 (1.4)
  FKSI-TSE; Month 9: number analyzed (Participants) | 26
  FKSI-TSE; Month 9 | 8.8 (2.7)
  FKSI-TSE; Month 12: number analyzed (Participants) | 16
  FKSI-TSE; Month 12 | 9.7 (2.7)
  FKSI-TSE; Month 18: number analyzed (Participants) | 11
  FKSI-TSE; Month 18 | 10.3 (1.4)
  FKSI-TSE; Month 24: number analyzed (Participants) | 5
  FKSI-TSE; Month 24 | 11 (1.2)
  FKSI-FWB; Day 0 | 6.3 (3.5)
  FKSI-FWB; Month 3: number analyzed (Participants) | 58
  FKSI-FWB; Month 3 | 5.0 (3.7)
  FKSI-FWB; Month 6: number analyzed (Participants) | 32
  FKSI-FWB; Month 6 | 6.3 (3.5)
  FKSI-FWB; Month 9: number analyzed (Participants) | 26
  FKSI-FWB; Month 9 | 5.8 (3.8)
  FKSI-FWB; Month 12: number analyzed (Participants) | 16
  FKSI-FWB; Month 12 | 6.4 (3.6)
  FKSI-FWB; Month 18: number analyzed (Participants) | 11
  FKSI-FWB; Month 18 | 5.9 (3.4)
  FKSI-FWB; Month 24: number analyzed (Participants) | 5
  FKSI-FWB; Month 24 | 5.2 (3.4)

ADVERSE EVENTS:
Time Frame: From date of sunitinib first dose until end of follow-up (up to maximum of 36 months)
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Sunitinib
All-Cause Mortality (participants affected / at risk) | 33/74
Serious Adverse Events (participants affected / at risk) | 35/74
Other Adverse Events (participants affected / at risk) | 35/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=74)
Death (General disorders) | 19
Pain (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Coma (Nervous system disorders) | 4
Hemorrhage intracranial (Nervous system disorders) | 2
Brain stem stroke (Nervous system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 2
Septic shock (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Hematuria (Renal and urinary disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 2
Circulatory collapse (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=74)
Diarrhea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucosal inflammation (General disorders) | 8
Asthenia (General disorders) | 4
Fatigue (General disorders) | 4
Pain (General disorders) | 2
Face oedema (General disorders) | 1
Inflammation (General disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Skin ulcer (Skin and subcutaneous tissue disorders) | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vision blurred (Eye disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Fungal infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03140176/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03140176/SAP_001.pdf